CLINICAL TRIAL: NCT04350567
Title: Role of the Metabotropic Glutamate Receptor Subtype 5 in Circadian Rhythm Misalignment and Depression: Implications for Treatment
Brief Title: Sleep/Wake Cycle and Depression: An Imaging and Treatment Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Christine DeLorenzo, Professor, Stony Brook University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1218123
Record Dates: First submitted 2020-03-17; First posted 2020-04-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-05

CONDITIONS: Depression; Major Depressive Disorder
MeSH Terms: conditions — Depression; Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental)
  Interventions: Other: Sleep Deprivation

INTERVENTIONS:
Other: Sleep Deprivation — On the first night, the participant sleeps normally as we assess their melatonin through blood work. On the second night, the participant has 3 PET/MRI scans. On the third night, the participant undergoes sleep deprivation. On the fourth night, the participant sleeps normally and we assess their melatonin again through blood work. Depression scores are taken before and after the intervention.

SUMMARY:
16.2 million American adults are affected by depression each year. The investigators are studying the relationship between sleep/wake cycle and depression. Mounting evidence suggests that abnormalities in circadian rhythms (biological changes that happen over the course of the day or night) are related to mood disorders. This may explain why people with depression frequently suffer with sleeping problems. The purpose of this study is to understand how circadian (sleep/wake) rhythms may be affected in depression and the best way to improve depression caused in this way. This will be performed by comparing circadian (sleep/wake) rhythms in people with and without depression.

The study involves being kept awake for one night. For depressed individuals, this technique will likely result in a brief (<1 day) improvement in depression. Following this study, participants with depression will be offered antidepressant medication at no cost. During the study, the investigators use brain scans to learn more about brain chemistry in health and depression.

DETAILED DESCRIPTION:
The study involves four overnight stays, three occurring consecutively and one occurring at a separate timepoint. For the three-night consecutive stay, on Overnight-1, sleep can occur as normal and the investigators will measure hormone levels during sleep. On Overnight-2, participants will be kept awake for around 36 hours. On Overnight-3, the investigators will measure hormone levels again during sleep. During a separately scheduled single overnight session (which happens sometime before or after the three-night consecutive stay), three sets of imaging over the course of the night are performed. The imaging is positron emission tomography (PET). It is designed to look at brain chemistry (particularly glutamate receptors in the brain). Participants may sleep in between scans. All participants with depression enrolled in the study will be seen by a clinician throughout the study and offered medication at no cost after the study.

Aim 1: Assess circadian (sleep/wake) phase in depressed and non-depressed individuals. Melatonin secretion is now an easily accessible circadian marker. Further, the average time interval between dim light melatonin onset (DLMO, the time at which melatonin rises above a certain threshold, "the most accurate biomarker of circadian phase position") and sleep midpoint (average bedtime plus half the average sleep duration) has been established as 6 hours in non-depressed participants and likely deviates from this optimum in major depressive disorder (MDD). For this reason, the investigators will measure melatonin in the blood on overnight visit 1.

Hypothesis 1. Average phase angle difference (DLMO - sleep midpoint) will be 6 hours (optimal) in healthy controls, but not depressed, participants.

Hypothesis 2. MDD severity (assessed by the Hamilton Depression Rating Scale, HDRS) will be correlated with deviation from optimal phase angle difference.

Aim 2: Assess brain chemistry (specifically one of the glutamate receptors, the metabotropic glutamate receptor subtype 5, mGluR5) expression at 3 times: the time of DLMO, peak and nadir of melatonin secretion (as measured from overnight visit 1). mGluR5 availability will be assessed near these times to capture mGluR5 circadian rhythmicity using PET and a tracer specific for mGluR5, [11C]ABP688.

Hypothesis 3. mGluR5 variation will be inverse to that of melatonin in both cohorts.

Aim 3: Determine the effect of acute sleep deprivation on circadian rhythms. Within approximately one week of Aims 1 & 2, all participants will receive sleep deprivation therapy. Following up to 36 hours of wakefulness (shown to increase mGluR5 at a single time point), the investigators will measure acute effects with repeat assessments of melatonin and depression severity. This will thus require two overnight stays in a row- one for the sleep deprivation and then the next to measure melatonin again in the blood while the participant sleeps.

Hypothesis 4. Sleep deprivation will be most successful in the depressed participants with greatest disruption in phase (Aim 1).

Hypothesis 5: Depressed participants will experience greater changes in phase angle difference following sleep deprivation than non-depressed participants.

Aim 4: To determine whether reliable estimates of [11C]ABP688 in plasma can be obtained using a miniPET scanner. [11C]ABP688 concentration will be measured at the wrist or leg with a novel synchronized PET scanner developed by Stony Brook Investigator, Dr. Paul Vaska. This innovative device provides estimates of plasma radioactivity simply by placing the participant's wrist or leg in a mini-PET scanner called versaPET. The radioactivity derived from this wrist or leg scanner, as well as the resulting outcome measures, will be compared to those estimated using blood analysis. This could make future PET studies easier by finding a substitute for blood sampling during the PET scan.

Uncovering the link between mGluR5, circadian disruption and MDD could:

(1) Identify biological underpinnings of circadian (sleep/wake) dysfunction; (2) Identify individuals (those with mGluR5 disruption) for whom treatments like sleep deprivation would be most effective; and (3) Increase use of this safe and rapid treatment.

ELIGIBILITY:
Inclusion criteria for depressed and non-depressed individuals

* Consent form signed
* Capacity to give informed consent
* Age 18 years or older (inclusive)
* Diagnosis of MDD and currently in a major depressive episode (depressed participants only)
* Score of at least twenty-nine on the MADRS (depressed participants only)

Exclusion Criteria:

* Participant considered at significant risk for suicide
* Unlikely to tolerate medication washout or the drug free period following washout (depressed participants only)
* Current psychosis
* ECT within 4 weeks of the first overnight visit
* Significant active physical illness or neurological deficit that may affect brain function or imaging
* A disease, job or life circumstance that creates an irregular circadian rhythm anticipated during the study
* Inability to maintain in bed and out of bed (regardless of sleep time, for depressed individuals) or sleep and wake times (for non-depressed individuals) to within ~30 min for a week before each overnight visit (will be measured by actigraphy and/or other measurements)
* Inability to abstain from medications that will affect glutamate levels or circadian rhythms, including stimulants, anti-epileptics, antidepressants, beta-blockers, hypnotics (including benzodiazepines), melatonin, or medications with glutamateric or GABAergic modes of action within 4 weeks before the first overnight visit as well as throughout the study
* Inability to reduce caffeine intake to <= ~300 mg of caffeine (~2.5 cups of coffee or equivalents) daily within 4 weeks of the first overnight visit as well as throughout the study
* Inability to abstain from nicotine within 4 weeks before the first overnight visit as well as throughout the study
* Inability to reduce use of alcohol to <= ~5 drinks per week from 4 weeks before the first overnight visit and throughout the study and to completely abstain from alcohol within 24 hours of any overnight visit
* Inability to abstain from significant substance use (including cannabis) within 4 weeks before the first overnight visit as well as throughout the study
* Planned intermittent fasting or calorie restricted diet within 4 weeks before the first overnight visit as well as throughout the study
* For females: Pregnancy within the past year, currently lactating; planning to conceive during the course of study participation, or abortion in the past two months
* Any MRI contraindications, including metal implants, pacemaker, metal prostheses, orthodontic appliances, or presence of shrapnel that are contraindicated for MRI
* Any PET contraindications, including if study imaging will result in the participant receiving greater exposure than the research limit, or if participant is currently breastfeeding

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Measure circadian phase in depressed and non-depressed individuals using the following outcome measure: phase angle difference (DLMO - sleep midpoint, units: hours) | 8 Weeks
  Hypothesis 1. Average phase angle difference (DLMO - sleep midpoint) will be 6 hours (optimal) in non-depressed participants. Hypothesis 2. MDD severity (assessed by the Hamilton Depression Rating Scale, HDRS) will be correlated with deviation from optimal phase angle difference. For this hypothesis, two outcome measures (phase angle difference, in hours) and HDRS (unitless, ranges from 0 to 52, higher numbers indicate worse depression severity) will be combined in the following way: the Pearson correlation coefficient will be assessed between the phase angle difference and HDRS of each individual. The correlation coefficient will be reported, and is expected to be positive.

SECONDARY OUTCOMES:
Measure mGluR5 expression (outcome measure: volume of distribution divided by free fraction) at the time of DLMO, peak and nadir of melatonin secretion. | 8 Weeks
  Hypothesis 3. mGluR5 variation will be inverse to that of melatonin in both cohorts. For this hypothesis, two outcome measures (mGluR5 expression at three time points) and (melatonin level at three time points) will be combined in the following way: the Pearson correlation coefficient will be assessed between mGluR5 expression and melatonin level within each individual. The correlation coefficient will be reported, and is expected to be negative.
Measure the effect of acute sleep deprivation on circadian rhythms (outcome measure: shift of the concentration of melatonin over time curve). | 8 Weeks
  Within approximately one week of Aims 1 & 2, all participants will receive sleep deprivation therapy. Following up to 36 hours of wakefulness (shown to increase mGluR5 at a single time point), we will measure acute effects with repeat assessments of melatonin. This will require two overnight stays in a row- one for the sleep deprivation and one to measure melatonin again in the blood while the participant sleeps.
To determine whether reliable estimates of [11C]ABP688 in plasma can be obtained using a miniPET scanner. | 8 Weeks
  Outcome measure: sum of square differences between [11C]ABP688 measured in blood samples compared to the concentration measured using the miniPET scanner.

CONTACTS AND LOCATIONS:
Locations (1):
- Stony Brook University Hospital, Stony Brook, New York, United States